CLINICAL TRIAL: NCT00324857
Title: Knee Replacement Disparity: A Randomized, Controlled Intervention
Brief Title: Educational Intervention for Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 05-234
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, Knee; race; ethnicity; knee replacement
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — Motivational Interviewing; Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1/Attention Control (Placebo Comparator): Subjects randomized to the attention control arm received a patient educational booklet about OA published by the National Institute of Arthritis and Musculoskeletal and Skin Diseases. This booklet provides a brief educational program that summarizes how to live with knee OA but does not specifically mention joint replacement
  Interventions: Other: Attention control
- Arm 2/Decision Aid (DA) (Active Comparator): Decision Aid Video: The research interventionist will show the participant the Dartmouth Knee OA Decision Aid video entitled "Treatment Choices for Knee Osteoarthritis." The video gives a detailed explanation of 1) the damage to the knee joint caused by OA; 2) treatment options including lifestyle changes, medications, injections, complementary therapy, and surgery; 3) the risks, benefits, and known efficacy of each treatment option.
  Interventions: Behavioral: Decision Aid Video
- Arm 3/ Motivational Interview (MI) (Active Comparator): Motivational Interviewing: The research intervention will conduct the fact-to-face MI session with the participant. This was used as a mechanism to help patients confront their thoughts about TKR and how to engage their primary care doctors about knee pain
  Interventions: Behavioral: Motivational Interviewing
- Arm 4/ DA and MI (Active Comparator): Decision Aid Video: The research interventionist will show the participant the Dartmouth Knee OA Decision Aid video entitled "Treatment Choices for Knee Osteoarthritis." The video gives a detailed explanation of 1) the damage to the knee joint caused by OA; 2) treatment options including lifestyle changes, medications, injections, complementary therapy, and surgery; 3) the risks, benefits, and known efficacy of each treatment option.
  Motivational Interviewing: The research intervention will conduct the fact-to-face MI session with the participant. This was used as a mechanism to help patients confront their thoughts about TKR and how to engage their primary care doctors about knee pain
  Interventions: Behavioral: MI plus Decision aid

INTERVENTIONS:
Behavioral: Decision Aid Video — The research interventionist will show the participant the Dartmouth Knee OA Decision Aid video entitled "Treatment Choices for Knee Osteoarthritis." The video gives a detailed explanation of 1) the damage to the knee joint caused by OA; 2) treatment options including lifestyle changes, medications, injections, complementary therapy, and surgery; 3) the risks, benefits, and known efficacy of each treatment option.
  Other Names: DA
  Arms: Arm 2/Decision Aid (DA)
Behavioral: Motivational Interviewing — The research intervention will conduct the fact-to-face MI session with the participant. The MI session will do the following things: 1) Assessing Readiness, Importance, and Confidence; 2) Eliciting Barriers, Concerns and Positive Motivational; 3) Summarizing Pros and Cons; 4) Assess Patient Values and Goals; 5) Provide a Menu of Options.
  Other Names: MI
  Arms: Arm 3/ Motivational Interview (MI)
Behavioral: MI plus Decision aid — Patient viewed the video and then underwent MI.
  Arms: Arm 4/ DA and MI
Other: Attention control — patients received a booklet.
  Arms: Arm 1/Attention Control

SUMMARY:
The purpose of this study is to demonstrate the efficacy of interventions to improve understanding of knee replacement risks, benefits, and expected outcomes among AA primary care patients, increase willingness to consider knee replacement among AA primary care patients, and increase primary care referral rates for surgical consideration for AA patients who meet the indications for knee replacement.

DETAILED DESCRIPTION:
The proposed project represents the next phase in a trajectory of VA research designed to eliminate racial disparities in the utilization of knee joint replacement - an effective treatment option for end-stage knee osteoarthritis (OA). Numerous studies have documented the existence of marked racial disparities in the utilization of knee joint replacement in OA. African-Americans (AA) are two to five times less likely than white patients to receive knee joint replacement for lower extremity OA. Our prior work has shown that compared to white patients, AA patients expect worse outcomes from this treatment and, consequently, are less willing to consider joint replacement even when clinically indicated and recommended by a physician. Patient willingness, an attitudinal disposition modifiable with education and counseling, has emerged as a key patient-level mediator in the utilization of elective medical procedures, such as knee joint replacement.

The short-term goals of this randomized, controlled trial are to demonstrate the efficacy of interventions to improve understanding of knee joint replacement risks, benefits, and expected outcomes among AA primary care patients, increase willingness to consider knee joint replacement among AA primary care patients, and increase primary care referral rates for surgical consideration for AA patients who meet the indications for knee joint replacement. We will test a multi-faceted intervention consisting of a knee OA decision aid video developed by the Foundation for Informed Medical Decision Making alone or in combination with individually tailored patient counseling using Motivational Interviewing versus an attention control. The long-term objective is to reduce or eliminate the racial gap in the utilization of knee joint replacement. The central hypothesis of this proposal is that the scientifically accurate, high quality patient-centered information on knee arthritis and joint replacement provided by the knee OA decision aid, alone or in combination with motivational interviewing, will improve patient understanding of knee joint replacement outcomes, increase patient willingness to consider knee joint replacement, and consequently lead to higher rates of referral for surgical consideration when clinically indicated. With increased referral rates, currently a major bottleneck in the path to joint replacement, more AA patients will receive recommendations for surgery, thus potentially reducing racial differences in the utilization of this procedure. This proposal is innovative because it is the first patient-centered evidence-based VA intervention trial to use a decision aid alone or in combination with motivational interviewing to intervene on a well-documented and marked racial disparity in joint replacement that exists within and outside the VA health care system.

Primary Specific Aims:

1. To examine the effectiveness of the proposed intervention strategies (DA alone, MI alone or a combined DA+MI)) to improve willingness to consider knee joint replacement when clinically indicated among AA primary care patients.
2. To examine the effectiveness of the proposed intervention strategies on patient expectations of knee joint replacement risks/benefits among AA primary care patients.
3. To examine the effectiveness of the proposed intervention strategies in increasing primary care referrals for surgical evaluation of AA patients with knee OA.

Secondary Specific Aim: To examine the effectiveness of the proposed intervention strategies to increase AA patient likelihood of receiving knee joint replacement within 12 months of the intervention.

A randomized, controlled factorial design will be utilized to examine the effectiveness of knee OA decision aid and/or MI compared with attention control on select key patient-centered and process of care outcomes. We will recruit approximately 600 AA primary care patients (150 at the VAPHS, 150 at the LSCDVAMC, and 300 at the PVAMC) who meet the American College of Rheumatology clinical indications for knee joint replacement and randomize them into either intervention arms or attention control. We will assess patient expectations, willingness and referral to joint replacement. We will also collect qualitative data on doctor-patient communication following the intervention or control so that we can assess (in the future) whether or not the interventions impact study outcomes through improved quality of communication. This study will provide hard evidence needed to improve quality of care for African-American VA patients who have end-stage knee OA, a major cause of disability and functional decline in VA elderly patients.

ELIGIBILITY:
Inclusion Criteria:

VA Pittsburgh Healthcare System, Philadelphia VA Medical Center, Louis Stokes Cleveland VAMC, AA primary care patients > age 50 who meet clinical criteria for knee OA (i.e., chronic, frequent knee pain based on the NHANES questions, WOMAC score = 39, and radiographic evidence of knee OA with K-L grade =2) are eligible for enrollment

Exclusion Criteria:

* Patients who have prior history of any:

  * major joint replacement
  * terminal illness (e.g., end-stage cancer)
  * physician-diagnosed inflammatory arthritis (i.e., rheumatoid arthritis, connective tissue disease, ankylosing spondylitis or other seronegative spondyloarthropathy)
  * contra-indications to replacement surgery (e.g., lower extremity paralysis as result of stroke)
* Patients who are not willing to be randomized
* Do not have the presence of knee OA
* Do not have telephone service

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 663 (Actual)
Dates: Start 2006-09; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Said A. Ibrahim, MD MPH, Principal Investigator — VA Medical Center, Philadelphia; C. Kent Kwoh, MD, Principal Investigator — University of Arizona
Locations (3):
- United States (3):
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA Medical Center, Philadelphia, Philadelphia, Pennsylvania
  - Division of General Medicine, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Ibrahim SA. Racial variations in the utilization of knee and hip joint replacement: an introduction and review of the most recent literature. Curr Orthop Pract. 2010 Mar;21(2):126-131. doi: 10.1097/BCO.0b013e3181d08223. PMID 21132110
- [Background] Emejuaiwe N, Jones AC, Ibrahim SA, Kwoh CK. Disparities in joint replacement utilization: a quality of care issue. Clin Exp Rheumatol. 2007 Nov-Dec;25(6 Suppl 47):44-9. PMID 18021506
- [Result] Ibrahim SA. Decision Aids and Elective Joint Replacement - How Knowledge Affects Utilization. N Engl J Med. 2017 Jun 29;376(26):2509-2511. doi: 10.1056/NEJMp1703432. No abstract available. PMID 28657869
- [Derived] Ibrahim SA, Hanusa BH, Hannon MJ, Kresevic D, Long J, Kent Kwoh C. Willingness and access to joint replacement among African American patients with knee osteoarthritis: a randomized, controlled intervention. Arthritis Rheum. 2013 May;65(5):1253-61. doi: 10.1002/art.37899. PMID 23613362

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1/Attention Control | Arm 2/Decision Aid (DA) | Arm 3/ Motivational Interview (MI) | Arm 4/ DA and MI
Started | 167 | 168 | 165 | 163
Completed | 161 | 162 | 158 | 158
Not Completed | 6 | 6 | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Arm 1/Attention Control: Attention control
- Arm 2/Decision Aid (DA): Decision Aid video
- Arm 3/ Motivational Interview (MI): Motivational Interviewing
- Arm 4/ DA and MI: Decision aid and MI
- Total: Total of all reporting groups
Arm/Group | Arm 1/Attention Control | Arm 2/Decision Aid (DA) | Arm 3/ Motivational Interview (MI) | Arm 4/ DA and MI | Total
Number analyzed (Participants) | 161 | 162 | 158 | 158 | 639
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (8) | 61 (9) | 61 (9) | 61 (8) | 61 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 161 | 162 | 158 | 158 | 639
Region of Enrollment [Number; unit: participants]
  United States | 161 | 162 | 158 | 158 | 639

OUTCOME MEASURES:

1. Primary Outcome: Change in Willingness.
Description: Change in willingness assessed using the willingness likert scale. The primary outcome was change in patient willingness to undergo total knee replacement. The willingness rating is a 5-category ordinal response scale from "definitely not willing" to "definitely willing" which was later dichotomized for analysis. Responses "definitely" and "probably willing" were combined and compared to "unsure", "probably not willing", and "definitely not willing" combined.
Time Frame: Follow-Up
Population: Study sample reflects the African American, predominantly male population of the VA health care system
Measure: Number; unit: participants
Arm/Group | Arm 1/Attention Control | Arm 2/Decision Aid (DA) | Arm 3/ Motivational Interview (MI) | Arm 4/ DA and MI
Number analyzed (Participants) | 161 | 162 | 158 | 158
participants
  1 Month Follow-Up | 1 | 1 | 1 | 1
  3 Month Follow-Up | 1 | 1 | 1 | 1
  12 Month Follow-Up | 1 | 1 | 1 | 1
Statistical Analysis 1: Comparison: Arm 1/Attention Control vs Arm 2/Decision Aid (DA) vs Arm 3/ Motivational Interview (MI) vs Arm 4/ DA and MI; Comparisons of the baseline demographic and clinical characteristics (TKR) across the 4 intervention groups were performed using chi-square tests for categorical data and analysis of variance for continuous variables. Willingness were compared across the groups over time using mixed-effect logistic regressions for dichotomous outcomes; Test type: Superiority or Other; p < 0.05, Regression, Logistic — Please note that although the outcome is measured using a Likert scale, for the analysis we dichotomized the results. P-value not adjusted for multiple comparison. Lastly, <0.05 is the actual computed P-value

2. Secondary Outcome: To Examine and Compare the Effectiveness of the Proposed Intervention Strategies to Increase AA Patient Likelihood of Receiving Knee Replacement Within 12 Months of the Intervention.
Time Frame: 12 months
Population: The data were not collected and therefore not analyzed.
Groups:
- Arm 4/ DA and MI: Decision Aid Video: The research interventionist will show the participant the Dartmouth Knee OA Decision Aid video entitled "Treatment Choices for Knee Osteoarthritis." The video gives a detailed explanation of 1) the damage to the knee joint caused by OA; 2) treatment options including lifestyle changes, medications, injections, complementary therapy, and surgery; 3) the risks, benefits, and known efficacy of each treatment option.
  Motivational Interviewing: The research intervention will conduct the fact-to-face MI session with the participant. This was used as a mechanism to help patients confront their thoughts about TKR and how to engage their primary care doctors about knee pain
  MI plus Decision aid: Patient viewed the video and then underwent MI.
Arm/Group | Arm 1/Attention Control | Arm 2/Decision Aid (DA) | Arm 3/ Motivational Interview (MI) | Arm 4/ DA and MI
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Arm 2/Decision Aid (DA): Decision Aid
Arm/Group | Arm 1/Attention Control | Arm 2/Decision Aid (DA) | Arm 3/ Motivational Interview (MI) | Arm 4/ DA and MI
Serious Adverse Events (participants affected / at risk) | 0/161 | 0/162 | 0/158 | 0/158
Other Adverse Events (participants affected / at risk) | 0/161 | 0/162 | 0/158 | 0/158

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes